CLINICAL TRIAL: NCT01470820
Title: Dose-response Relationship of Phototherapy for Hyperbilirubinaemia Using Diodes: is There a "Saturation Point"?
Brief Title: Dose-response Relationship of Phototherapy for Hyperbilirubinaemia Using Diodes: is There a "Saturation Point"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: N-20090014
Record Dates: First submitted 2011-11-04; First posted 2011-11-11 (Estimated); Last update posted 2011-11-11 (Estimated); Status verified 2011-11

CONDITIONS: Neonatal Hyperbilirubinemia
Keywords: Neonates; Hyperbilirubinemia; Phototherapy; Light irradiance; Saturation point
MeSH Terms: conditions — Hyperbilirubinemia, Neonatal; Hyperbilirubinemia | interventions — Phototherapy; Blue Light

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Distance 20 cm (Active Comparator): The infants were randomized by sealed and opaque envelopes to one of four phototherapy regimens. Either with distance from the phototherapy device to the mattress of 20, 29, 38 or 47 cm measured by a wood stick for each infant, corresponding to the distances to the infants of averagely 12, 21, 30 and 39 cm, respectively.
  Interventions: Other: Phototherapy with blue light
- Distance 29 cm (Active Comparator)
  Interventions: Other: Phototherapy with blue light
- Distance 38 cm (Active Comparator)
  Interventions: Other: Phototherapy with blue light
- Distance 47 cm (Active Comparator)
  Interventions: Other: Phototherapy with blue light

INTERVENTIONS:
Other: Phototherapy with blue light — The infants were placed in a bassinet with the phototherapy device placed above them. All infants were exposed naked (apart from eye pads and diaper) to continuously phototherapy for 24 hours, interrupted only for feeding and nursing for 30 minutes every three hours. TsB was determined before phototherapy and after 24 hours of treatment. The phototherapy apparatus used was neoBLUE LED phototherapy device (Natus Medical Inc., San Carlos, CA, USA) emitting blue light with an emission peak at 460 nm and a bandwidth of 450-470 nm. The irradiance was measured by use of the neoBLUE LED phototherapy radiometer (Natus Medical Inc.) every 8th hour at the infants head, trunk and knees and the average was calculated. The radiometer measures spectral irradiance in the range 420-500 nm with maximum sensitivity in the spectrum 440-480 nm.

SUMMARY:
Background: Using light emitting diodes (LED's) during conventional phototherapy it is possible to reduce the distance from light source to infant, thereby increasing light irradiance.

Objective: To examine the relation between light irradiance and the rate of decrease in total serum bilirubin concentration (TsB) and to see if the investigators can identify a "saturation point", i.e. an irradiation level above which there is no further decrease in TsB.

Design: Prospective randomised study. Setting: Neonatal Intensive Care Unit, Pediatric Department, Aalborg Hospital, Aarhus University Hospital, Denmark.

Material and method: 151 infants with gestational age ≥ 33 weeks and uncomplicated hyperbilirubinaemia are randomised to one of 4 different distances from phototherapy device to mattress (20, 29, 38 and 47 cm). TsB is measured before and after 24 hours of phototherapy and irradiance every 8th hour. Main outcome measure is 24 hours decrease of TsB expressed in percent (∆ TsB0-24 (%)).

ELIGIBILITY:
Inclusion Criteria:

* Gestational age ≥ 33 weeks
* Uncomplicated neonatal hyperbilirubinemia

Exclusion Criteria:

* < 33 weeks
* infants in incubators

Min Age: 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-07; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
24 hours decrease of TsB expressed in percent. | Baseline and 24 hours
  TsB was measured before and after 24 hours of phototherapy and irradiance every 8th hour. Main outcome was 24 hours decrease of TsB expressed in percent (∆ TsB0-24(%).

CONTACTS AND LOCATIONS:
Overall Officials: Pernille K Vandborg, MD, Principal Investigator — Pediatric department, Aalborg Sygehus, Aarhus University Hospital; Finn Ebbesen, Professor, Principal Investigator — Pediatric department, Aalborg Sygehus, Aarhus University Hospital
Locations (1):
- Pediatric Department, Aalborg Sygehus, Aarhus University Hospital, Aalborg, Denmark

REFERENCES:
- [Derived] Vandborg PK, Hansen BM, Greisen G, Ebbesen F. Dose-response relationship of phototherapy for hyperbilirubinemia. Pediatrics. 2012 Aug;130(2):e352-7. doi: 10.1542/peds.2011-3235. Epub 2012 Jul 16. PMID 22802603